CLINICAL TRIAL: NCT03600116
Title: Collection of Breath and Sweat to Identify Indicators of Hypoglycemia
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mitre Medical Corp. (Industry)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2018P000868
Record Dates: First submitted 2018-06-19; First posted 2018-07-26 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breath and sweat samples will be collected and shipped to the collaborator, the MITRE Corporation, for analysis. Blood samples will be collected to measure plasma glucose, but will be discarded after the measurement is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Visit: After consent and enrollment, subjects with type 1 diabetes will arrive to the study visit having fasted the night before. Subjects will be given a meal, and will be given an insulin injection for this meal, calculated based on their prescribed meal to carbohydrate ratio as well as a correction bolus to correct their current plasma glucose value down to 40 mg/dL based on their prescribed insulin sensitivity factor. Following the insulin injection, subjects will eat breakfast and be observed in the clinic setting. Blood, breath, and sweat samples will be collected throughout the study visit with increased frequency of collection during hypoglycemia. After subjects reach the hypoglycemia threshold, they will be allowed to eat and drink and their blood sugar will be monitored for stability prior to discharge.

SUMMARY:
Subjects with type 1 diabetes will be observed in the diabetes research center clinic following a meal and an insulin injection. Breath and sweat samples will be collected at intervals throughout the visit, with increased frequency during hypoglycemia. Collaborators with the MITRE Corporation will perform analyses on these samples to identify any relationships between volatile organic compounds in breath and sweat and hypoglycemia.

DETAILED DESCRIPTION:
Subjects enrolled in the study will have clinical type 1 diabetes managed with rapid acting insulin. After consent and enrollment, they will arrive to the study visit having fasted the night before. Subjects will be given a meal, and will be given an insulin injection for this meal, calculated based on their prescribed meal to carbohydrate ratio as well as a correction bolus to correct their current plasma glucose value down to 40 mg/dL based on their prescribed insulin sensitivity factor. Following the insulin injection, subjects will eat breakfast and be observed in the clinic setting. Blood, breath, and sweat samples will be collected throughout the study visit with increased frequency of collection during hypoglycemia. Collaborators with the MITRE Corporation will perform analyses on these samples to identify any relationships between volatile organic compounds in breath and sweat and hypoglycemia. After subjects reach the hypoglycemia threshold, they will be allowed to eat and drink and their blood sugar will be monitored for stability prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the subject documented prior to any study procedures
* Age ≥ 18 years
* Have had clinical type 1 diabetes for at least one year
* Willing and able to avoid deodorant, scented lotions, and scented laundry detergent on your clothes on the day of the visit

Exclusion Criteria:

* Unable to provide informed consent (e.g. impaired cognition or judgment)
* Unable to safely comply with study procedures and reporting requirements (e.g. impaired memory or unable to speak and read English)
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception

  * Subjects must use acceptable contraception for the two weeks prior to the study, throughout the study and for the two weeks following the study.
  * Acceptable contraception methods include:
  * Oral contraceptive pill (OCP)
  * Intrauterine Device (IUD, hormonal or copper)
  * Male condoms
  * Female condoms
  * Diaphragm or cervical cap with spermicide
  * Contraceptive patch (such as OrthoEvra)
  * Contraceptive implant (such as Implanon, Nexplanon)
  * Vaginal ring (such as NuvaRing)
  * Progestin shot (such as Depo-Provera)
  * Male partner with a vasectomy proven to be effective by semen analysis
* Abnormal EKG consistent with coronary artery disease or increased risk of malignant arrhythmia including, but not limited to, evidence of active ischemia, prior myocardial infarction, proximal LAD critical stenosis (Wellen's sign), prolonged QT interval (> 440 ms). Non-specific ST segment and T wave changes are not grounds for exclusion in the absence of symptoms or history of heart disease. A reassuring evaluation by a cardiologist after an abnormal EKG finding may allow participation.
* History of hypoglycemic seizures (grand mal) or coma in the last year
* History of poor venous access or inadequate venous access as determined by trial nurse or physician at time of screening
* Hemoglobin < 12 g/dl for men, < 11 g/dl for women
* Any factors that, in the opinion of the principal investigator would interfere with the safe completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers who fit the selection criteria will be considered as candidates for this study. The study team will contact individuals who have previously inquired about participation in our studies and have asked to have their contact information kept on file. In addition, advertisements for the study may be posted at the MGH Diabetes Center and other places, and may be distributed in the weekly broadcast email of research studies seeking volunteers. A letter may be sent to adult endocrinologists in the Boston metropolitan as well as selected nearby endocrinologists informing them of the study and asking them to refer any eligible patients who might be interested.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Identification of Volatile Organic Chemical Indicators of Hypoglycemia | Up to 12 months
  Exploration via chemical analysis of clinical samples taken from diabetics' breath and sweat, using gas chromatograph-mass spectrometry (GC-MS) and liquid chromatograph-mass spectrometry (LC-MS), to determine the volatile organic compounds whose varying concentrations might correlate with diabetics' blood sugar concentrations in the normoglycemic and hypoglycemic ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital (MGH) Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The study data may be shared with collaborators at the MITRE Corporation (a non-profit research corporation), but only in a form in which all personally identifiable information has been removed. Shared data will be in the form of a database in which only a number identifies subjects.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03600116/Prot_SAP_000.pdf